CLINICAL TRIAL: NCT01564121
Title: Phase 2 Study of the Effect of Zoledronate on Local Recurrence After Surgical Treatment of Giant Cell Tumors of Bone
Brief Title: Study of the Effect of Zoledronate on Local Recurrence After Surgical Treatment of Giant Cell Tumors of Bone Zométa
Acronym: Zometa
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/10-E
Record Dates: First submitted 2011-06-28; First posted 2012-03-27 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Giant Cell Tumors of Bone
MeSH Terms: interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: acid Zoledronic — Treatment with zoledronic acid will be initiated during hospitalization, the day after the removal of redundant. Intravenous injection of 4 mg. of zoledronate diluted in sodium chloride 9 / 1000 or a solution of 5% dextrose in intravenous over 15 minutes. In the absence of intolerance clinic, an infusion of zoledronic acid in the same doses and modalities will be performed in a hospital (on the occasion of a follow-up visit after surgery) at the 3rd, 6th, 9th and 12th weeks after the first, or 5 injections. )

SUMMARY:
The giant cell tumor (GTC) is an aggressive benign bone tumor, growing at the metaphyseal-epiphyseal regions of long bones, especially around the knee and the distal radius.It is responsible for bony destruction in para-articular zone fracture and leading to the breakdown and destruction of the underlying joint.

Histologically, the tumor cell contains a contingent of monocytic cells round, a contingent of giant type cell of type osteoclastic responsible for bone resorption that accompanies these tumors and a contingent of lengthened cells fibroblast-like considered to be contingent tumor.

The treatment is exclusively surgical; or by resection of the lesion which takes away tumour and its environment, solution which, if it prevents local recurrence, imposes an important bony and articular reconstruction, always limited and deteriorating rapidly over time in these young patients; or by curettage of lesion, by "hollowing-out" of the bone, creating a hole which it will be necessary to fill up by a bony grafting or a substitute of the bone (cement). This last solution, if it preserves a better function, exposes at risk of local recurrence,putting into play the prognosis of articulation near, most often the knee.Despite different local adjuvants treatments used during surgical operation, after having curetted the cavity and before filling it up, the recidivism rates vary from 12 % to 41 % (average 25 %) in literature.

The beneficial effect of the adjuvants therapeutics suggests the concept broadly accepted by a tumoral microscopic residual at the origin of the local recidivism .Biphosphonates (BP) is molecules which settle in vivo on the hydroxyapatite of the bone; they inhibit the recruitment of the osteoclast forerunners and the activity of mature osteoclast. Besides, biphosphonates containing some nitrogen (N-BP), leads to the apoptose of mature osteoclast. These molecules also have a direct effect on tumor cells , causing apoptosis of neoplastic cells of myeloma, of breast cancer. Clinical controlled studies confirm the experimental data of N-BP. Two work also showed their effect on osteoclasts and stroma cells of tumours with giant cells but no clinical study assessed potential on the prevention of the local recurrence.

The investigators offer a study phase 2 of the effectiveness of N-BP (acid zoledronique) on the prevention of the local recurrence of tumours with primary huge cells after surgical treatment by curettage - filing by a surgeon referent in oncologic orthopedic surgery.

Number of patients: 24

DETAILED DESCRIPTION:
Outcome Measures:

- Main: occurrence of recurrence detectable by Reasonable Magnetic Imaging (IRM) and / or standardized radiography.

Local recurrence will be discussed in the presence or appearance on the radiographic and IRM monitoring of an osteolysis in the periphery of the cavity curetted, does not exist on the radio in post-operative with IRM signal abnormalities in the same location,taking the gadolinium. If in doubt, a new surgical biopsy will confirm or not the diagnosis of local recurrence

secondary:

* clinical: patient interview, clinical examination
* biological Complete blood count, creatinine, serum calcium, phosphate, magnesium

ELIGIBILITY:
Inclusion Criteria:

* Patient age (18 years)
* Benign giant cell tumor of the bone histologically confirmed after biopsy
* Non-metastatic tumor
* The first surgical treatment of the tumor
* Indication of conservative treatment with curettage, filling asked by the surgeon investigator
* Written consent of the patient

Exclusion Criteria:

* Minor patient
* Location of a pulmonary TCG
* Surgical indication of prior or immediately en bloc resection
* Need for treatment with an aminoglycoside
* Against-indication for zoledronic acid: pregnancy, lactation, known hypersensitivity to this drug or another bisphosphonate, severe renal impairment or a previous kidney failure, severe bradycardia or conduction disturbance on ECG.
* Dental Problems in progress, including an infection of the teeth or jaw underlying (mandible and maxilla), dental trauma or recent diagnosis or history of osteo-necrosis of the jaw (ONJ) , or exposure of the OSE or delayed healing after dental procedures.
* Dental or jaw bone recent (within 6 weeks) or planned (extractions, implants, ...).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Decrease in the recurrence rate of GTC of the bone after surgery (efficacy). | 36 months

SECONDARY OUTCOMES:
Tolerance at the filling treatment with zoledronic acid (safety). | 36 months
  Clinical examination of the patient, clinical examination (confusing yes / no, headache yes / no, visual yes / no, nausea yes / no, vomiting yes / no, itching rash yes / no, arthralgia yes / no, bone pain yes / no, bradycardia <60 during the infusion yes / no, fever yes / no, taste thirst yes / no, chest pain yes / no)
  * Organic: blood count (NFS), creatinine, serum calcium, phosphate, magnesium (below the standards of the laboratory that conducted the review yes / no)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France